CLINICAL TRIAL: NCT01202448
Title: Prospective Cohort Study With Risk-adapted Central Nervous System Evaluation in Diffuse Large B-cell Lymphoma
Brief Title: Prospective Cohort Study With Central Nervous System Evaluation in Diffuse Large B-cell Lymphoma
Acronym: PROCESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Asan Medical Center (Other); Yonsei University (Other); National Cancer Center, Korea (Other Government); Korea Cancer Center Hospital (Other); Korea University (Other)
Responsible Party: Principal Investigator, Kim, Seok Jin, Associate professor, Samsung Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010-04-091
Record Dates: First submitted 2010-09-08; First posted 2010-09-15 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Diffuse large B cell lymphoma; central nervous system; prognosis
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DLBCL with risk factor (Active Comparator): Patients have any of risk factors for secondary CNS involvement
  Interventions: Procedure: CSF analysis

INTERVENTIONS:
Procedure: CSF analysis — The cerebrospinal fluid will be evaluated via lumbar puncture.
  Other Names: Brain MRI

SUMMARY:
This study is to evaluate the incidence of central nervous system (CNS) relapse or metastasis in patients with diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
We dichotomize patients according to the risk of CNS involvement. Then, we perform CNS evaluation in patients at risk of CNS involvement. We prospectively monitor whether CNS relapse or metastasis occurs in patients with diffuse large B-cell lymphoma

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed patients with diffuse large B cell lymphoma
2. > 20 years
3. life expectancy more than 6 months
4. Written informed consent

Exclusion Criteria:

1. Refusal to informed consent
2. Lymphomas other than diffuse large B cell lymphoma
3. Primary CNS lymphoma

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2010-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
CNS relapse/involvement | Up to 2 years after participants are enrolled.
  After enrollment, patients will be monitored to check the CNS relapse or involvement

SECONDARY OUTCOMES:
survival | Up to 2 years after participants are enrolled
  The survival outcome of patients will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Cheolwon Suh, MD, PhD, Principal Investigator — Consortium for Improving Survival of Lymphoma
Locations (2):
- South Korea (2):
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul